CLINICAL TRIAL: NCT05193006
Title: Assessment of Histologic Prognostic Factors in Peritoneal Malignant Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1120
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Peritoneal Malignant Mesothelioma
Keywords: prognostic factors; peritoneal malignant mesothelioma; mesothelioma
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- peritoneal malignant mesothelioma of grade 1: peritoneal malignant mesothelioma of grade 1
  Interventions: Other: No intervention
- peritoneal malignant mesothelioma of grade 2: peritoneal malignant mesothelioma of grade 2
  Interventions: Other: No intervention
- peritoneal malignant mesothelioma of grade 3: peritoneal malignant mesothelioma of grade 3
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Malignant peritoneal mesothelioma is a rare neoplasm. The most common type, the epithelioid type, has been further divided into histological patterns of tubulo-papillary, acinar, adenomatoid, micropapillary, or solid. Its prognosis is improved by the use of a locoregional treatment combining extensive cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC), which increases survival up to 50 months. Histology is one of the most important prognostic variable that, forms the basis for treatment decisions. However, the prognostic of the epithelioid type varies greatly due to its tumor heterogeneity. It is therefore necessary to find prognostic factors of malignant epithelioid peritoneal mesothelioma in order to better define the therapeutic strategy. Among histological factors, solid growth, tumor necrosis, nuclear atypia, and mitotic count were found to be independent prognostic factors in epithelioid malignant pleural mesothelioma. However, in epithelioid malignant peritoneal mesothelioma (EMPM), these factors were studied in small and heterogeneous series in terms of histological growth and definitions used for histological factors. The present large study was conducted to investigate the prognostic impact of several histologic factors in EMPM. Their prognosis impacts were assessed using overall survival (OS) and progression-free survival (PFS) in EMPM.

ELIGIBILITY:
Inclusion Criteria:

* - peritoneal malignant mesothelioma

Exclusion Criteria:

* opposition to reuse personnal data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: squamous cell carcinoma of the oropharynx
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of pronostic impact of nuclear grade in comparison with combined grade in peritoneal malignant mesothelioma | 3 months to 4 years
  Assessment by the review of pathologists

CONTACTS AND LOCATIONS:
Locations (6):
- UZ Gent, Ghent, Belgium
- University Hospital of Lyon, Pierre-Bénite, France
- Institut f. Pathologie und Neuropathologie, Tübingen, Germany
- Zydus Hospitals, Ahmedabad, India
- The Norwegian Radium Hospital, Oslo, Norway
- Fundação Champalimaud, Lisbon, Portugal